CLINICAL TRIAL: NCT03249103
Title: A Phase 2, Single-Blind, Exploratory, Placebo-controlled, Pilot Study to Assess the Efficacy and Safety of Daily Oral NYX-2925 in Subjects With Fibromyalgia
Brief Title: Evaluate the Efficacy and Safety of NYX-2925 in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aptinyx (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYX-2925-2002
Record Dates: First submitted 2017-08-02; First posted 2017-08-15 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — NYX-2925

STUDY DESIGN:
Intervention Model Description: All subjects will receive placebo, NYX-2925 20 mg QD, NYX-2925 200 mg QD for sequential 2 week treatment periods, then go into Follow-up for 1 week.
Masking Description: Subjects are masked to the sequence in which they are taking placebo QD, NYX-2925 20 mg QD, NYX-2925 200 mg QD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All subjects (Experimental): Up to 24 subjects will receive placebo, NYX-2925 20 mg QD, and NYX-2925 200 mg QD for sequential 2 week treatment periods, then go into Follow-up for 1 week.
  Interventions: Drug: NYX-2925; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: NYX-2925 — NYX-2925 is a novel small molecule that modulates the N-methyl-D-aspartate receptor (NMDAR).
Drug: Placebo oral capsule — Matching placebo capsules.

SUMMARY:
The primary objective is to determine whether daily dosing with NYX-2925 changes markers of central pain processing in subjects with fibromyalgia by evaluating changes in evoked pain, and visual stimulation, functional magnetic resonance imaging (fMRI), resting state function connectivity magnetic resonance imaging (rs-fcMRI) and proton magnetic resonance spectroscopy (H-MRS) in fibromyalgia subjects on active drug versus placebo.

DETAILED DESCRIPTION:
This is a single-blind, exploratory, placebo-controlled, pilot study to assess the efficacy and safety of daily oral NYX-2925 in fibromyalgia subjects. The study will include a screening period (up to 30 days), a placebo period, an active treatment period with, and a follow-up period as follows:

* Placebo PO Every Day (QD) for 2 weeks
* NYX-2925 PO QD for 2 weeks (2x)
* Follow-up for 1 week

Eligible subjects will receive MRIs during the screening period, during the placebo period, during the NYX-2925 PO QD period. Safety assessments will be conducted and adverse events will be collected during the study. Daily pain scores and other fibromyalgia scales will be collected during the study. Daily pain scores and other fibromyalgia scales will be collected for exploratory analysis. During the follow-up period, an optional MRI will be completed for consenting subjects in order to evaluate duration of effect.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects meets the 2010 American College of Rheumatology (ACR) criteria for fibromyalgia.
2. Self-reported clinical pain ≥ 4 and on the Numeric Pain Rating Scale (NPRS) at screening and baseline.
3. Subject receives and agrees to remain on their stable fibromyalgia treatment plan established at least 14 days prior to dosing.
4. Subject agrees to use only non-steroidal anti-inflammatory (NSAID) or acetaminophen treatment as needed for breakthrough pain, and/or, zopiclone, zolpidem, zaleplon, or eszopiclone for sleep (if needed).
5. Right handed.
6. Calculates creatinine clearance ≥ 60 mL/minute.
7. Female subjects of child bearing potential with a negative serum pregnancy test prior to entry into the study and who are practicing an adequate method of birth control (e.g., surgical sterilization, oral or parenteral contraceptives, intrauterine device that is considered safe for MRI procedures, barrier [condom with spermicide]) and who do not plan to become pregnant, breastfeed, or donate ova during the course of the study and for 28 days after the final administration of investigational product.
8. Ability to understand the requirements of the study, provide written informed consent, abide by the study restrictions, and agree to return for the required assessments.

Exclusion Criteria:

1. Current or expected use of opioid or narcotic analgesics, monoamine oxidase inhibitors (MAOIs), tricyclic antidepressants, gabapentins, topiramate, anticonvulsants, benzodiazepines, and sedatives, or hypnotics.
2. Unstable doses of allowed antidepressants or muscle relaxants. Use of NSAIDs or acetaminophen 24 hours prior to imaging procedures is prohibited.
3. Pain due to concurrent disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, or other chronic widespread pain condition(s) that may confound fibromyalgia pain.
4. Untreated endocrine disorder that may confound fibromyalgia assessments.
5. Psychiatric or cognitive disorder (e.g., current schizophrenia, severe depression, suicidal ideation, dementia, etc.).
6. Clinically significant alcohol or other substance abuse within the last 2 years.
7. Positive screen for medically inappropriate or illegal use of drugs of abuse.
8. Current treatment with medications such as ketamine, amantadine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
9. History of allergy, sensitivity, or intolerance to medications such as ketamine, amantadine, dextromethorphan, memantine, methadone, dextropropoxyphene, or ketobemidone.
10. Women, who are pregnant, breast feeding, or planning to become pregnant or donate ova during the course of the study and for 28 days after the final administration of investigational product.
11. Huntington's, Parkinson's, Alzheimer's, Multiple Sclerosis, or history of seizures, epilepsy, or strokes.
12. Contraindications to fMRI procedures. These may include but are not limited to: surgical clips, surgical staples, metal implants, and certain metallic dental material.
13. Current or habitual use (within the last 12 months) of artificial nails, nails enhancements, or nail extensions that cover any portion of either thumbnail.
14. Abnormal laboratory results, medical history, or concurrent conditions that would preclude safe study participation, or interfere with study procedures/assessments.
15. Impaired liver function.
16. Known history of significant heart condition or high blood pressure.
17. Current evidence of dysplasia or history of cancer malignancy (including lymphoma and leukemia) in the last 5 years.
18. Human immunodeficiency virus (HIV) infection, hepatitis, or other ongoing infectious disease.
19. History of severe kidney or liver impairment.
20. History of migraine.
21. History of lower limb vascular surgery or current lower limb vascular dysfunction.
22. Received an investigational drug or device within 30 days of dosing.
23. Previous treatment with NYX-2925.
24. Resting heart rate < 45 or ≥ 95 beats per minute.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Aptinyx Clinical Site, Ann Arbor, Michigan
  - Aptinyx Clinical Site, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Approximately 24 subjects were planned to be enrolled. Twenty-two (22) subjects were enrolled.
Groups:
- All Treated Subjects: Subjects received Placebo, 20 mg NYX-2925 once daily (QD), and 200 mg NYX-2925 QD
Period: Overall Study
Arm/Group | All Treated Subjects
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- All Treated Subjects: Subjects received Placebo, 20 mg NYX-2925 QD, and 200 mg NYX-2925 QD
Arm/Group | All Treated Subjects
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (15.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Fibromyalgia disease history, years [Mean (Standard Deviation); unit: years] | 14.57 (14.476)

OUTCOME MEASURES:

1. Primary Outcome: Mean (SD) Glx/Total Creatine Levels in Dorsal Anterior Cingulate Cortex (dACC): NYX-2925 20 mg and 200 mg PO QD at Week 4 and Week 6, Respectively.
Time Frame: Week 2, Week 4, Week 6
Population: Population includes study subjects with analyzable images (n=20)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Treated Subjects
Number analyzed (Participants) | 20
ratio
  dACC mean placebo | 2.1670 (0.17796)
  dACC mean NYX-2925 20 mg | 2.0550 (0.19710)
  dACC NYX-2925 200 mg | 2.0975 (0.19141)
Statistical Analysis 1: Comparison: All Treated Subjects; placebo - NYX-2925 20 mg; Test type: Other; p = 0.032, t-test, 2 sided

2. Primary Outcome: Mean (SD) Changes in Posterior Insula (pINS) Glx/Total Creatine Levels Before and After Acute Painful Pressure Stimulation: NYX-2925 20 mg and 200 mg PO QD at Week 4 and Week 6, Respectively.
Time Frame: Week 2, Week 4, and Week 6
Population: Population includes study subjects with analyzable images (n=19)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | All Treated Subjects
Number analyzed (Participants) | 19
ratio
  pINS mean placebo | 1.993 (0.13981)
  pINS mean NYX-2925 20 mg | 1.911 (0.14242)
  pINS NYX-2925 200 mg | 1.903 (0.16194)
Statistical Analysis 1: Comparison: All Treated Subjects; placebo - NYX-2925 200 mg; Test type: Other; p = 0.039, t-test, 2 sided

3. Other Pre Specified Outcome: Mean Change in Numeric Pain Rating Scale (NPRS) Score Assessing Average Pain in the Past 24 Hours
Description: Numeric pain rating scale is a unidimensional segmented numeric version of the visual analog scale. A subject selects a whole number (0 to 10) that best indicates the intensity of their pain, where 0 represents no pain and 10 the worst pain imaginable.
Time Frame: Change from Baseline, Week 2 (Placebo), Week 4, and Week 6 (NYX-2925)
Population: The efficacy population is based on subjects included in the safety population and have at least one post-baseline visit after receiving NYX-2925 20 mg PO QD.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Treated Subjects
Number analyzed (Participants) | 18
units on a scale
  Baseline | 5.32 (1.411)
  Week 2 | 4.82 (1.275)
  Week 4 | 4.74 (1.360)
  Week 6 | 4.12 (1.650)
Statistical Analysis 1: Comparison: All Treated Subjects; Test type: Other; p = 0.0072, t-test, 2 sided; comparing Week 2 (Placebo) to Week 6 (NYX-2925 200 mg)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the informed consent was signed to the end of the subject's participation in the study (Week 7).
Description: Adverse Events were collected and are summarized for all NYX-2925 exposure. Adverse events were not collected with regard to specific dose.
Groups:
- All Treated Subjects: Subjects received Placebo, 20 mg NYX-2925 QD, and 200 mg NYX-2925 QD. Adverse Events were collected and are summarized for all NYX-2925 exposure. Adverse events were not collected with regard to specific dose.
Arm/Group | All Treated Subjects
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 7/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Treated Subjects (N=22)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Diarrhoea/ (Gastrointestinal disorders) | 2 (2)
Eructation (Gastrointestinal disorders) | 2 (2)
Tension headache (Nervous system disorders) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT03249103/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT03249103/SAP_001.pdf